CLINICAL TRIAL: NCT02047513
Title: Neoadjuvant Plus Adjuvant or Only Adjuvant Nab-Paclitaxel Plus Gemcitabine for Resectable Pancreatic Cancer: A Prospective, Randomized, Controlled, Phase II Study of the AIO (Working Group for Medical Oncology From the German Cancer Society) Pancreatic Cancer Group
Brief Title: Neoadjuvant Plus Adjuvant or Only Adjuvant Nab- Paclitaxel Plus Gemcitabine for Resectable Pancreatic Cancer
Acronym: NEONAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Celgene (Industry); ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-PAK-0313; 2013-005559-34 (EudraCT Number); AX_CL_PANC_AIO_003710 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2014-01-09; First posted 2014-01-28 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Resectable Pancreatic Cancer; Ductal Adenocarcinoma of the Pancreas
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- perioperative nab-paclitaxel/gemcitabine (Experimental): neoadjuvant chemotherapy (8 weeks) preceding surgery (3 weeks after completion of chemotherapy) followed by adjuvant chemotherapy (16 weeks, begin within 12 weeks after surgery)
  Interventions: Drug: perioperative nab-paclitaxel/gemcitabine
- adjuvant nab-paclitaxel/gemcitabine (Experimental): Surgery followed by adjuvant chemotherapy (24 weeks, begin within 12 weeks after surgery), follow-up per patient: Until end of study or death
  Interventions: Drug: adjuvant nab-paclitaxel/gemcitabine

INTERVENTIONS:
Drug: perioperative nab-paclitaxel/gemcitabine — 2 cycles of nab-paclitaxel/gemcitabine (nab-paclitaxel 125 mg/m2, gemcitabine 1000 mg/m2 on day 1, 8 and 15 of an 28 day-cycles) followed by 3 weeks of rest and subsequent tumor surgery. Starting within 12 weeks after surgery adjuvant chemotherapy with 4 cycles of nab-paclitaxel/gemcitabine (nab-paclitaxel 125 mg/m2, gemcitabine 1000 mg/m2 on day 1, 8 and 15 of an 28 day-cycles)
  Arms: perioperative nab-paclitaxel/gemcitabine
Drug: adjuvant nab-paclitaxel/gemcitabine — Tumor surgery followed by adjuvant chemotherapy with 6 cycles of nab-paclitaxel/gemcitabine (nab-paclitaxel 125 mg/m2, gemcitabine 1000 mg/m2 on day 1, 8 and 15 of an 28 day-cycles, starting within 12 weeks after surgery)
  Arms: adjuvant nab-paclitaxel/gemcitabine

SUMMARY:
NEONAX is an interventional, prospective, randomized, controlled, open label, two sided survival phase II studies against a fixed survival probability, with an unconnected analysis of the results in both experimental arms.

Determining the impact of 2 cycles of Perioperative nab-paclitaxel/gemcitabine followed by surgery and 4 cycles of adjuvant nab-paclitaxel/gemcitabine or 6 cycles of adjuvant nab-paclitaxel/gemcitabine on the Disease free survival (DFS) rate at 18 months post randomization

DETAILED DESCRIPTION:
The planned trial will enable us to address the following issues:

* Identification of patients who benefit from surgery. Tumor progress during intensified Perioperative chemotherapy is likely to indicate a particularly poor prognosis suggesting that these patients would not have benefitted from immediate surgery.
* Assess tumor response/downsizing using nab-paclitaxel/gemcitabine also at the molecular level
* Can we achieve a better systemic tumor control or reduce the metastatic spread using nab-paclitaxel/gemcitabine compared to adjuvant gemcitabine
* Examining the effect of a more efficacious chemotherapy regimen (nab-paclitaxel/gemcitabine) in the adjuvant setting
* Defining the impact of a perioperative or adjuvant chemotherapy with gemcitabine/nab-paclitaxel on DFS and 3-year Overall survival (OS)

Histopathological tumor regression will be evaluated in addition to tumor size measurement according to Response Evaluation Criteria In Solid Tumors (RECIST). We will establish a histopathological tumor regression score to evaluate the efficacy of the neoadjuvant treatment. For this score we will examine tumor core biopsies obtained prior to neoadjuvant treatment and histological tumor specimen after surgery in both arms.

To reliably determine R0 resections, the resected specimen will be prepared for pathology in a defined manner according to the procedure set out in the German S3 guidelines for pancreatic cancer.

This trial provides the unique opportunity in pancreatic cancer to obtain material prior to and after surgery for biomarker analysis and correlation with outcome. We will perform pharmacogenomic candidate gene analysis of hENT1 (human equilibrative nucleoside transporter-1), CDA (cell differentiation agent), DCK (Desoxycytidin-Kinase) and 5´nucleotidase in both arms.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytological confirmed, clearly resectable ductal adenocarcinoma of the pancreas (PDAC) ≤ cT3 with no prior tumor specific treatment.
* No evidence of metastases to distant organs (e.g. liver, peritoneum, lung).
* Resectable tumor. Determination of resectability based on spiral CT scans with both oral and i.v. contrast enhancement or on MRI using a recent consensus definition (Resectability: Clear fat planes around the celiac artery, hepatic artery and superior mesenteric artery.)
* Measurable tumor according to RECIST 1.1
* ECOG performance status 0 or 1
* Creatinine clearance ≥ 30 ml/min
* Serum total bilirubin level ≤ 2.5 x ULN (not necessary for enrollment or randomization, but before start of neoadjuvant chemotherapy in arm A)
* ALT and AST ≤ 2.5 x ULN (not necessary for enrollment or randomization, but before start of neoadjuvant chemotherapy in arm A)
* In case of biliary obstruction, biliary decompression is required if the patient was randomized to receive neoadjuvant chemotherapy (arm A)
* White blood cell count ≥ 3.5 x 106/ml, neutrophil granulocytes count ≥ 1,5 x 106/ml, platelet count ≥ 100 x 106/ml
* Signed informed consent incl. participation in translational research
* Age ≥ 18 years

Exclusion criteria:

* Borderline resectable PDAC by radiologic criteria
* Papillary cancer
* Neuroendocrine Cancer
* Tumor specific pre-treatment
* Local recurrence
* Peritoneal or other distant metastases
* Radiographic evidence of severe portal hypertension/cavernous transformation
* Infiltration of extrapancreatic organs (except duodenum)
* Ascites
* Gastric outlet obstruction
* Global respiratory insufficiency requiring oxygen supplementation
* Chronic infectious diseases, immune deficiency syndromes
* Premalignant hematologic disorders, e.g. myelodysplastic syndrome
* Disability to understand and sign written informed consent document
* Past or current history of malignancies except for the indication under this study and curatively treated:

  * Basal and squamous cell carcinoma of the skin
  * In-situ carcinoma of the cervix
  * Other malignant disease without recurrence after at least 2 years of follow-up
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment
* Clinically relevant or history of interstitial lung disease, e.g. non-infectious pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan or chest x-ray.
* History of or evidence upon physical examination of CNS disease unless adequately treated (e.g. primary brain tumor, seizure not controlled with standard medical therapy or history of stroke).
* Pre-existing neuropathy > grade 1 (NCI CTCAE)
* Allogeneic transplantation requiring immunosuppressive therapy or other major immunosuppressive therapy
* Severe non-healing wounds, ulcers or bone fractions
* Evidence of bleeding diathesis or coagulopathy
* Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and PTT < 1.5 ULN within 28 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution)
* Major surgical procedures, except open biopsy, nor significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgical procedure during the course of the study except for surgery of pancreatic cancer with curative intent and central intravenous line placement for chemotherapy administration.
* Pregnancy or breastfeeding women.
* Subjects with known allergies to the study drugs or to any of its excipients.
* Current or recent (within the 28 days prior randomization) treatment with another investigational drug or participation in another investigational study.
* Any psychological, familial, sociological or geographical condition potentially compromising compliance with the study protocol and the follow-up schedule; those conditions should be discussed with the patient prior to registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Time to Disease free survival (DFS) | 18 months after randomization
  To improve the DFS rate at 18 months in at least one arm to≥ 55%

SECONDARY OUTCOMES:
Safety | 57 months
  • Safety of nab-paclitaxel/gemcitabine in the neoadjuvant and adjuvant setting
morbidity and mortality | 7 years
  • pre- and postoperative morbidity and mortality in both studies
toxicity | 57 months
  • Dropout rate due to toxicity in the neoadjuvant study
Disease progression | 7 years
  • Disease progression during neoadjuvant therapy
resection rate | 53 months
  • R0 and R1 resection rate in both groups as assessed according to the German S3 guidelines
Tumor response | 57 months
  • Tumor response according to RECIST v1.1; histopathological regression based on a predefined pathological handling of the resected specimen in the perioperative study
Correlation of tumor regression and R0 resection | 57 months
  • Correlation of tumor regression and R0 resection rate with response according to RECIST v1.1 in the perioperative study
Overall survival | 7 years
  • Overall survival in both studies
tumor recurrence | 7 years
  • First site of tumor recurrence in both studies
quality of life | 57 months
  • Explorative analysis of health related quality of life in both studies
pharmacogenomic markers, tumor-biomarkers and molecular analyses | 57 months
  • Correlation of DFS, OS and tumor regression with pharmacogenomic markers, tumor-biomarkers and molecular analyses in both studies
Safety | 57 months
  • Assessment of safety
Tumor response | 66 months
  To assess tumor response using the imaging data (CT scans, MRI-scans) obtained during the trial
Tumor recurrence | 66 months
  To assess tumor recurrence using the imaging data (CT scans, MRI-scans) obtained during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, Prof. Dr., Principal Investigator — University of Ulm, Dept. of Internal Medicine I
Locations (1):
- University of Ulm, Dept. of Internal Medicine I, Ulm, Germany

REFERENCES:
- [Derived] Seufferlein T, Uhl W, Kornmann M, Algul H, Friess H, Konig A, Ghadimi M, Gallmeier E, Bartsch DK, Lutz MP, Metzger R, Wille K, Gerdes B, Schimanski CC, Graupe F, Kunzmann V, Klein I, Geissler M, Staib L, Waldschmidt D, Bruns C, Wittel U, Fichtner-Feigl S, Daum S, Hinke A, Blome L, Tannapfel A, Kleger A, Berger AW, Kestler AMR, Schuhbaur JS, Perkhofer L, Tempero M, Reinacher-Schick AC, Ettrich TJ. Perioperative or only adjuvant gemcitabine plus nab-paclitaxel for resectable pancreatic cancer (NEONAX)-a randomized phase II trial of the AIO pancreatic cancer group. Ann Oncol. 2023 Jan;34(1):91-100. doi: 10.1016/j.annonc.2022.09.161. Epub 2022 Oct 7. PMID 36209981
- [Derived] Ettrich TJ, Berger AW, Perkhofer L, Daum S, Konig A, Dickhut A, Wittel U, Wille K, Geissler M, Algul H, Gallmeier E, Atzpodien J, Kornmann M, Muche R, Prasnikar N, Tannapfel A, Reinacher-Schick A, Uhl W, Seufferlein T. Neoadjuvant plus adjuvant or only adjuvant nab-paclitaxel plus gemcitabine for resectable pancreatic cancer - the NEONAX trial (AIO-PAK-0313), a prospective, randomized, controlled, phase II study of the AIO pancreatic cancer group. BMC Cancer. 2018 Dec 29;18(1):1298. doi: 10.1186/s12885-018-5183-y. PMID 30594153
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de